CLINICAL TRIAL: NCT04643301
Title: Liraglutide for Low-responders After Bariatric Surgery
Acronym: LIBAR
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Cancellation by sponsor
Sponsor: Zuyderland Medisch Centrum (Other)
Collaborators: Nederlandse Obesitas Kliniek (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NOK0020
Record Dates: First submitted 2020-11-02; First posted 2020-11-25 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Obesity; Obesity, Morbid
Keywords: Obesity; Liraglutide; GLP-1; Bariatric Surgery; Weight loss; Low-responders
MeSH Terms: conditions — Obesity; Obesity, Morbid; Weight Loss | interventions — Liraglutide

STUDY DESIGN:
Intervention Model Description: The study cohort will be compared to a retrospective matched cohort based on BMI before surgery, gender and type of surgery
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adding Liraglutide to current treatment program (Experimental): Adding 3,0mg of Liraglutide to the current treatment program of low-responders 3 months after bariatric surgery.
  Interventions: Drug: Liraglutide Pen Injector

INTERVENTIONS:
Drug: Liraglutide Pen Injector — Daily subcutaneous injection of 3.0mg liraglutide (GLP-1 antagonist) for low-responders 3 months after bariatric surgery.
  Other Names: Saxenda

SUMMARY:
To study the effect of Liraglutide (3.0 mg daily) on 9-month weight loss in low responders 3-months after bariatric surgery.

DETAILED DESCRIPTION:
Rationale: In 20 - 30% of the patients sufficient weight loss is not achieved (low responders) after bariatric surgery. Secondary and/or tertiary bariatric procedures can lead to successful weight loss and resolution of comorbid conditions though, morbidity and mortality rates of these procedures are high. Therefore, additional pharmacotherapy has been suggested. Liraglutide is one of the medications that might improve outcome in the post-bariatric population. It is a Glucagon-like peptide-1 receptor analogue developed to treat type 2 diabetes which causes glucose-dependent insulin secretion and promotes satiety and inhibits glucagon secretion. In obese (non-bariatric) patients, Liraglutide has shown to improve glycemic control, decrease blood pressure, lower cardiovascular risk and decrease body weight. There are only a few small retrospective trials assessing the effect of additional pharmacotherapy in low responders after bariatric surgery. These trials show promising results, with weight loss up to 9.7 % and limited side-effects.

Objective: To study the effect of Liraglutide (3.0 mg daily) on 9-month weight loss in low responders 3-months after bariatric surgery.

Study design: Pragmatic trial.

Study population: Bariatric patients with a pre-operative BMI ≥ 35.0 kg/m2 who have undergone a primary Roux-en-Y gastric bypass or sleeve gastrectomy, are treated with group consultations by the Nederlandse Obesitas Kliniek and are low responders at 3-months follow-up for which they will be treated with the plus module. A low responder is defined by comparing the measured percentage total weight loss (%TWL) at the 3-month follow-up with the expected weight loss. When %TWL is below the 25% quartile of expected weight loss the patient is considered a low responder. The plus module is an extra intervention our clinic provides for the patients who are considered low responders at the 3-month follow-up moment after surgery, this is part of our standard care program.

Intervention: Addition of Liraglutide 3.0 mg daily for 6 months to standard care.

Main study parameters/endpoints: The primary objective is to study the effect of Liraglutide (3.0 mg daily) on 9-month weight loss in low responders after bariatric surgery. The secondary objectives are the description of persistence of therapy and used daily dose, gastro-intestinal symptoms and eating habits and weight loss up to 36 months after surgery.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The burden of participation consists of extra usage of medication which patients have to administer subcutaneously daily, the extra consultations and two questionnaires. The risks consist of the mainly gastro-intestinal side-effects.

ELIGIBILITY:
Inclusion Criteria:

* BMI before surgery was ≥ 35.0 kg/m2
* Patient is treated with group consultation at the NOK
* Patient has undergone a primary Roux-en-Y gastric bypass (RYGB) or sleeve gastrectomy (SG)
* Patient is in the lowest %TWL quartile, 3 months after surgery and will be enrolled in the plus module.

Exclusion Criteria:

* Type 1 or type 2 diabetes
* Decreased renal function (creatinine clearance < 30 ml/min)
* Liver failure (all)
* Congestive heart failure or angina pectoris NYHA class III and IV
* Malignancy in history
* Pancreatitis (in history)
* Pregnancy / breast-feeding
* Inflammatory Bowel Disease
* Thyroid malignancy in history
* Use of warfarin or other coumarin derivates

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12-21 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
%TWL (%TWL) | 6 months
  To study of the effect of six months treatment with Liraglutide (3.0 mg daily) on 9-month weight loss (%TWL) in low responders after bariatric surgery.

SECONDARY OUTCOMES:
Persistence | 6 months
  To describe the persistence of therapy. Number and percentage of patients who are able to tolerate the treatment throughout the study.
GI symptoms | 6 months
  To describe the gastro-intestinal symptoms of the study group. Gastro-intestinal symptoms and eating habits of the patients will be assessed in two ways, first by adverse event rapportage and second with the "eating habits and physical problems" scales of the BODY-Q questionnaire (see F1 questionnaire) which will be administered at study start and at 14 weeks after study start.
%TWL | 12, 18, 24 and 36 months
  To study the weight change at 12, 18, 24 and 36 months after surgery
Dosage in mg | 6 months
  To describe the average daily dose patients use:
  * Number and percentage of patients in whom dose escalation was according to protocol.
  * Number and percentage of patients who used 3.0 mg as a daily dose for 22 weeks.
  * Average daily dose of all patients (after the dose escalation)
Eating habits | 6 months
  To describe the eating habits of the study group. Gastro-intestinal symptoms and eating habits of the patients will be assessed in two ways, first by adverse event rapportage and second with the "eating habits and physical problems" scales of the BODY-Q questionnaire (see F1 questionnaire) which will be administered at study start and at 14 weeks after study start.

CONTACTS AND LOCATIONS:
Overall Officials: J.W. Greve, MD, PHD, Principal Investigator — Nederlandse Obesitas Kliniek/Zuyderland Medisch Centrum

IPD SHARING:
Plan to Share IPD: Undecided